CLINICAL TRIAL: NCT02475317
Title: A Randomized, Blinded, Placebo-controlled, Phase 1 Study to Assess the Relative Potency of Multiple Oral Doses of LUM001 and SHP626 in Overweight and Obese Adult Subjects, as Assessed by Fecal Bile Acid Excretion
Brief Title: Study to Assess the Relative Potency of Multiple Oral Doses of LUM001 and SHP626 in Overweight and Obese Adults as Assessed by Fecal Bile Acid Excretion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SHP625-101
Record Dates: First submitted 2015-06-10; First posted 2015-06-18 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Healthy Volunteers
Keywords: Volunteer
MeSH Terms: interventions — maralixibat; volixibat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Placebo (Placebo Comparator): Participants will receive placebo matched to maralixibat 10 milligram (mg), 20 mg, 50 mg once daily (QD), 50 mg twice daily (BID), 100 mg liquid formulation and volixibat 10 mg, 20 mg capsule orally for 7 days.
  Interventions: Drug: Placebo
- Maralixibat 10mg (Experimental): Participants will receive maralixibat 10 mg liquid formulation orally QD for 7 days.
  Interventions: Drug: Maralixibat
- Volixibat 10mg (Experimental): Participants will receive volixibat 10 mg capsule orally QD for 7 days.
  Interventions: Drug: Volixibat
- Maralixibat 20mg (Experimental): Participants will receive maralixibat 20 mg liquid formulation orally QD for 7 days.
  Interventions: Drug: Maralixibat
- Volixibat 20mg (Experimental): Participants will receive volixibat 20 mg capsule orally QD for 7 days.
  Interventions: Drug: Volixibat
- Maralixibat 50mg (Experimental): Participants will receive maralixibat 50 mg liquid formulation orally QD for 7 days.
  Interventions: Drug: Maralixibat
- Maralixibat 50mg BID (Experimental): Participants will receive maralixibat 50 mg liquid formulation orally BID for 7 days.
  Interventions: Drug: Maralixibat
- Maralixibat 100mg (Experimental): Participants will receive maralixibat 100 mg liquid formulation orally QD for 7 days.
  Interventions: Drug: Maralixibat

INTERVENTIONS:
Drug: Placebo — Participants will receive placebo matched to maralixibat/volixibat orally for 7 days.
  Arms: Placebo
Drug: Maralixibat — Participants will receive maralixibat in 10 mg, 20 mg, 50 mg or 100 mg doses.
  Other Names: LUM001
  Arms: Maralixibat 100mg; Maralixibat 10mg; Maralixibat 20mg; Maralixibat 50mg; Maralixibat 50mg BID
Drug: Volixibat — Participants will receive volixibat in 10 mg and 20 mg doses.
  Other Names: SHP626
  Arms: Volixibat 10mg; Volixibat 20mg

SUMMARY:
The purpose of this study is to assess the relative potency of multiple oral doses of LUM001 and SHP626 administered for 7 days as assessed by fecal bile acid excretion in overweight and obese adult subjects. This study is designed to address the relative potency question for the first time in the same.

ELIGIBILITY:
Inclusion Criteria:

1. An understanding, ability, and willingness to fully comply with study procedures, study diet, and restrictions.
2. Ability to voluntarily provide written, signed, and dated (personally or via a legally-authorized representative) informed consent/and assent as applicable to participate in the study.
3. Aged 18-65 years inclusive at the time of consent. The date of signature of the informed consent is defined as the beginning of the screening period. This inclusion criterion will only be assessed at the first screening visit.
4. Males who agree to comply with any applicable contraceptive requirements of the protocol or females of non-childbearing potential (see Section 4.4 for details).
5. Must be considered generally healthy. Health status is defined by the absence of evidence of any active or chronic disease (see Section 7.2.2.1 for details and exceptions) following the completion of a detailed medical and surgical history, a complete physical examination, vital signs, 12-lead ECG, hematology, blood chemistry, and urinalysis.
6. Must have a body mass index of 25.0-35.0 kg/m² inclusive with a body weight >63.5 kg (140 lbs at the first screening visit). This inclusion criterion will only be assessed at the first screening visit.
7. All clinical laboratory parameters are within normal laboratory limit or not found to be clinically significant by the principal investigator.
8. Ability to swallow a dose(s) of investigational product(s).

Exclusion Criteria:

1. History of any hematological, hepatic, respiratory, cardiovascular, renal, neurological, or psychiatric disease, gall bladder removal, or current or recurrent disease that could affect the action, absorption, or disposition of the investigational product, or clinical or laboratory assessments.
2. Current or relevant history of physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully complete the study, or any condition that presents undue risk from the investigational product or procedures.
3. Known or suspected intolerance or hypersensitivity to the investigational product(s), closely-related compounds, or any of the stated ingredients.
4. Significant illness, as judged by the investigator, within 2 weeks prior to the first dose of investigational product.
5. Known history of alcohol or other substance abuse within the last year.
6. Donation of blood or blood products (eg, plasma or platelets) within 60 days prior to receiving the first dose of investigational product.
7. Within 30 days prior to the first dose of investigational product:

   * Have used an investigational product (if elimination half-life is <6 days, otherwise 5 half-lives).
   * Have been enrolled in a clinical study (including vaccine studies) that, in the investigator's opinion, may impact this Shire-sponsored study.
   * Have had any substantial changes in eating habits or exercise routine, as assessed by the investigator
8. Confirmed resting systolic blood pressure >145 mmHg or <89 mmHg, and diastolic blood pressure >95 mmHg or <59 mmHg.
9. Twelve-lead ECG demonstrating QTc >460 milliseconds for male subjects or >470 milliseconds for female subjects at screening. If QTc exceeds 460 milliseconds for males or 470 milliseconds for females, the ECG should be repeated 2 more times and the average of the 3 QTc values should be used to determine the subject's eligibility
10. A positive screen for drugs of abuse at screening or at Day -3 (check-in).
11. Male subjects who consume more than 21 units of alcohol per week or 3 units per day. Female subjects who consume more than 14 units of alcohol per week or 2 units per day. (1 alcohol unit=1 beer or 1 wine [5 oz/150 mL] or 1 liquor [1.5 oz/40 mL] or 0.75 oz alcohol).
12. A positive HIV, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody screen.
13. Use of tobacco (eg, smoking or chewing) or other nicotine-containing products (eg, gum, patch) in any form. Ex-users must report that they have stopped using tobacco for at least 30 days prior to receiving the first dose of investigational product.
14. Routine consumption of more than 2 units of caffeine per day or subjects who experience caffeine withdrawal headaches. (One caffeine unit is contained in the following items: one 6 oz [180 mL] cup of coffee, two 12 oz [360 mL] cans of cola, one 12 oz cup of tea, and three 1 oz [85 g] chocolate bars. Decaffeinated coffee, tea, and cola are not considered to contain caffeine.)
15. Prior screen failure, randomization, participation, or enrollment in this study. If a subject has successfully completed a study using LUM001 or SHP626, they may participate in this study providing at least 30 days has passed since their last dose of these investigational products and they have successfully completed all screening procedures
16. Current use of any medication (including over-the-counter, herbal, or homeopathic preparations) with the exception of those medications listed in Section 5.2.1. (Current use is defined as use within 14 days of the first dose of investigational product.)
17. An inability to follow a standardized diet and meal schedule or inability to fast, as required during the study.
18. Colonoscopy, barium enema, or other tests that require a bowel cleansing within 4 weeks prior to the first dose of investigational product.
19. Subjects who report typically having less than 3 bowel movements per week or greater than 3 bowel movements per day.
20. Use of antibiotics within 30 days prior to the first dose of investigational product.
21. Use of bile acid sequestrants within 30 days prior to the first dose of investigational product

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-06-01; Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
Change From Baseline of Fecal Bile Acid Excretion After Dosing (Day 6 and Day 7) | Baseline, Day 7
  Fecal bile acid excretion was determined by the concentration of total bile acids in stool samples over each 24-hour collection window during the lead-in and treatment periods.

SECONDARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Baseline up to follow-up (up to 16 days)
  An adverse event is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An AE (classified by preferred term) that occurred during the treatment period was considered a TEAE if it had a start date on or after the first dose of IMP; it had a start date before the date of the first dose of IMP, but increased in severity on or after the date of the first dose of the blinded IMP.
Change From Baseline in Vital Signs (Supine Pulse Rate and Standing Pulse Rate) at Day 8 / End of Treatment (ET) | Baseline, Day 8
  Supine Pulse Rate and Standing Pulse Rate were reported.
Change From Baseline in Vital Signs (Blood Pressure) at Day 8 / End of Treatment (EOT) | Baseline, Day 8
  Supine Systolic Blood Pressure (Supine SBP); Standing Systolic Blood Pressure (Standing SBP); Supine Diastolic Blood Pressure (Supine DBP); Standing Diastolic Blood Pressure (Standing DBP) were reported.
Change From Baseline in 12-lead Electrocardiogram (ECG) - Heart Rate at Day 8 / End of Treatment (EOT) | Baseline, Day 8
  Twelve-lead ECG was performed.
Change From Baseline in 12-lead ECG Intervals at Day 8 | Baseline, Day 8
  Twelve-lead ECG was performed. The corrected QT interval (QTc) was derived by Bazett formula (QTcB=QT/(RR)^1/2) and Fridericia formula (QTcF=QT/(RR)^1/3). PR Interval; QRS Interval; QT Interval; QTcB Interval; QTcF Interval, RR Intervals were reported.
Number of Participants with Clinically Meaningful Changes in Serum Biochemistry Laboratory Parameters | Baseline up to Day 8
  Number of participants with clinically meaningful changes in serum biochemistry laboratory parameters were reported.
Number of Participants with Clinically Meaningful Changes in Coagulation and Hematology Parameters | Baseline up to Day 8
  Activated partial thromboplastin time (aPTT), hematocrit, hemoglobin, monocytes and erythrocytes were analyzed. Number of participants with clinically meaningful change in coagulation and hematology parameters were reported.
Number of Participants With Clinically Meaningful Changes in Urinalysis Parameters | Baseline up to Day 8
  Number of participants with clinically meaningful changes in urinalysis parameters were reported.
Change From Baseline in Total Serum Bile Acid Concentration at Day 7 | Baseline, Day 7
  Serum bile acid concentrations were determined using a validated liquid chromatography with tandem mass spectrometric detection (LC/MS/MS) method.
Change From Baseline in Serum Concentration of 7- alpha-hydroxy-4-cholesten-3-one (C4) at Day 7 | Baseline, Day 7
  Serum samples were assayed for C4 using a validated LC/MS/MS method.
Stool Hardness Measured by Bristol Stool Chart at Day 7 | Day 7
  Stool hardness was assessed according to the Bristol Stool Chart, where 1 was the hardest and 7 was the softest form of stool. Types 3 and 4 were considered normal and types at either end of the scale were considered severe.
Frequency of Bowel Movements at Day 7 | Day 7
  Frequency of bowel movements were calculated by treatment group and by day.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Mirum
Locations (1):
- New Orleans Center for Clinical Research, Knoxville, Tennessee, United States